CLINICAL TRIAL: NCT06940856
Title: The Impact of Chloride Imbalance on BPD Development and Mortality in Preterm Infants
Brief Title: Chloride Imbalance in Preterm Infants
Status: Not yet recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Murat Köstü, Neonatologist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Murat Kostu
Record Dates: First submitted 2025-04-07; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Bronchopulmonary Dysplasia (BPD); Mortality Prediction; Chloride Disorder
Keywords: Bronchopulmonary dysplasia; Preterm infant; Mortality; Chloride imbalance
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — YSH1 protein, S cerevisiae

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Infants without dyschloremia: Infants with serum chloride levels within reference range before 36 weeks PMA
  Interventions: Other: Incomplete response; Other: Complete response; Other: Bad response
- Infants with dyschloremia: Infants with serum chloride levels <96 mEq/l and >110 mEq/l before 36 weeks PMA
  Interventions: Other: Incomplete response; Other: Complete response; Other: Bad response

INTERVENTIONS:
Other: Incomplete response — Infants died before 36 weeks PMA, infants diagnosed to have BPD at 36 weeks PMA and infants developed major complications before 36 weeks PMA:
  1. >Stage 2 necrotizing enterocolitis according to Bell classification
  2. Hemodynamically significant patent ductus arteriosus
  3. >Grade 2 intraventricular hemorrhage,
  4. Retinopathy of prematurity, ICROP classification stage >2
  5. >Stage 2 cystic periventricular leukomalacia
  6. Ventricular dilatation/hydrocephalus requiring intervention
Other: Complete response — Infants discharged before 36 weeks PMA and infants who reached 36 weeks PMA without BPD and major complications:
  1. >Stage 2 necrotizing enterocolitis according to Bell classification
  2. Hemodynamically significant patent ductus arteriosus
  3. >Grade 2 intraventricular hemorrhage,
  4. Retinopathy of prematurity, ICROP classification stage >2
  5. >Stage 2 cystic periventricular leukomalacia
  6. Ventricular dilatation/hydrocephalus requiring intervention
Other: Bad response — Infants died before 36 weeks PMA and infants diagnosed to have BPD at 36 weeks PMA

SUMMARY:
In adults and children low or high blood chloride levels are linked to the risk of death. The aim of this observational study is to determine whether there is a relationship between low or high blood chloride levels and the risk of death or long-term lung problems. We will also learn the risk factors and associated conditions of high or low blood chloride levels. We will include infants born before 32 weeks of pregnancy or have a birth weight of less than 1500 grams in the study. The main question it aims to answer is:

Is there a relationship between low or high blood chloride levels in the first 4-6 weeks of life and risk of death or long-term lung problems in premature babies? We will examine the medical reports of babies who were followed up in neonatal intensive care unit over the past 5 years.

DETAILED DESCRIPTION:
Chloride balance usually parallels that of sodium, and it is strictly correlated to the extracellular volume balance. In addition plasma chloride and bicarbonate concentrations are inversely regulated through the chloride-bicarbonate exchange pump in renal collecting ducts, independent of sodium. Consequently, plasma chloride levels are closely correlated with pH (hypochloremia/metabolic alkalosis, hyperchloremia/metabolic acidosis).

In adults, dyschloremia is associated with mortality, acute kidney injury, and prolonged hospital stay. Hyperchloremia is often associated with severe sepsis. It has been shown that resuscitation with high-chloride fluids (eg: saline solution) instead of balanced fluids (e.g., Ringer's lactate) increases the need for inotropes in critically ill adults. Similarly, hyperchloremia in septic pediatric patients is linked to acute renal injury requiring dialysis, increased inotropic support, and mortality. In 1979, infants fed with chloride-deficient formula were reported to develop impaired head growth and neurologic sequelae.

Although serum chloride is routinely measured in neonatal intensive care units, its clinical significance is often overlooked. For this reason unlike sodium, literature on chloride metabolism in preterm infants is exceedingly limited.

Advancements in perinatal care over the past 50 years have significantly improved survival rates in preterm infants. However, a large proportion of very preterm infants who survive the neonatal period develop bronchopulmonary dysplasia (BPD). BPD, a chronic lung disease, manifests clinically through persistent respiratory support and/or oxygen dependency. Despite efforts to optimize neonatal care -such as controlled oxygen usage, non-invasive ventilation, volume-guarantee techniques, high-frequency ventilation, and caffeine therapy- BPD remains the most common complication among preterm infants and is associated with increased morbidity and mortality.

It has been suggested that extracellular volume expansion (edema) plays a role in the pathophysiology of BPD. Perlman et al.'s 1986 study demonstrated that infants who died from BPD exhibited hypochloremia, metabolic alkalosis, and complications like inadequate head growth, more frequently than those who survived. These findings highlight the critical importance of chloride imbalance in neonates, similar to findings in adult and pediatric populations.

This study aims to investigate the relationship between chloride balance and two major outcomes-mortality and the development of BPD-in preterm infants. Infants <32 weeks postmentruel age (PMA) or weighing less than 1500 grams will be enrolled in the study. We also plan to explore the relationship of dyschloremia with other outcomes of prematurity (eg: patent ductus arteriosus, ventilator dependency, retinopathy of prematurity (ROP), necrotizing enterocolitis, intraventricular hemorrhage, periventricular leukomalacia, hospital stay. Lastly we plan to explore the risk factors and clinical/laboratory conditions that are associated with chloride level abnormalities.

If this study yields findings that underscore the clinical significance of chloride levels in preterm infants, similar to adults and children, then close monitoring of chloride balance and appropriate interventions could potentially reduce mortality and BPD incidence in preterm infants. Conversely, if results indicate that chloride balance lacks clinical significance in preterm infants, this will also contribute valuable information to the current literature.

ELIGIBILITY:
Inclusion Criteria:

* Infants born <32 weeks PMA or <1500 grams
* Infants admitted to NICU within the first 24 hours

Exclusion Criteria:

* Infants with major congenital anomalies
* Infants with chromosomal anomalies
* Infants who have undergone enterostomy operation
* Infants admitted to NICU after the first 24 hours

Ages: 1 Hour to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population includes infants admitted to the Neonatal Intensive Care Unit at Kanuni Sultan Suleyman Training and Research Hospital over the past 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
BPD | From enrollment to the end of 36 weeks PMA
  BPD at 36 weeks PMA

SECONDARY OUTCOMES:
Mortality | From enrollment to the end of 36 weeks PMA
  Mortality within 36 weeks PMA

OTHER OUTCOMES:
NEC | From enrollment to the end of 36 weeks PMA
  >Stage 2 necrotizing enterocolitis according to Bell classification within 36 weeks PMA
PDA | From enrollment to the end of 36 weeks PMA
  Hemodynamically significant patent ductus arteriosus within 36 weeks PMA
IVH | From enrollment to the end of 36 weeks PMA
  >Grade 2 intraventricular hemorrhage within 36 weeks PMA
ROP | From enrollment to the end of 36 weeks PMA
  Retinopathy of prematurity, ICROP classification stage >2 at 36 weeks PMA
PVL | From enrollment to the end of 36 weeks PMA
  >Stage 2 cystic periventricular leukomalacia at 36 weeks PMA
Hydrocephalus | From enrollment to the end of 36 weeks PMA
  Ventricular dilatation/hydrocephalus requiring intervention at 36 weeks PMA

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Education and Research Hospital, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We are not sure that local ethics committee that approved our study will allow IPD sharing

REFERENCES:
- [Background] Perlman JM, Moore V, Siegel MJ, Dawson J. Is chloride depletion an important contributing cause of death in infants with bronchopulmonary dysplasia? Pediatrics. 1986 Feb;77(2):212-6. PMID 2935779
- [Background] Thebaud B, Goss KN, Laughon M, Whitsett JA, Abman SH, Steinhorn RH, Aschner JL, Davis PG, McGrath-Morrow SA, Soll RF, Jobe AH. Bronchopulmonary dysplasia. Nat Rev Dis Primers. 2019 Nov 14;5(1):78. doi: 10.1038/s41572-019-0127-7. PMID 31727986
- [Background] Chutorian AM, LaScala CP, Ores CN, Nass R. Cerebral dysfunction following infantile dietary chloride deficiency. Pediatr Neurol. 1985 Nov-Dec;1(6):335-41. doi: 10.1016/0887-8994(85)90067-0. PMID 3880419
- [Background] Khan AH, Gai J, Faruque F, Bost JE, Patel AK, Pollack MM. Pediatric Mortality and Acute Kidney Injury Are Associated with Chloride Abnormalities in Intensive Care Units in the United States: A Multicenter Observational Study. J Pediatr Intensive Care. 2020 Nov 23;11(2):91-99. doi: 10.1055/s-0040-1719172. eCollection 2022 Jun. PMID 35734213
- [Background] Kalikkot Thekkeveedu R, Ramarao S, Dankhara N, Alur P. Hypochloremia Secondary to Diuretics in Preterm Infants: Should Clinicians Pay Close Attention? Glob Pediatr Health. 2021 Feb 4;8:2333794X21991014. doi: 10.1177/2333794X21991014. eCollection 2021. PMID 33614850
- [Background] Iacobelli S, Kermorvant-Duchemin E, Bonsante F, Lapillonne A, Gouyon JB. Chloride Balance in Preterm Infants during the First Week of Life. Int J Pediatr. 2012;2012:931597. doi: 10.1155/2012/931597. Epub 2012 Mar 8. PMID 22505945